CLINICAL TRIAL: NCT01088646
Title: Evaluation of PillCam® Express Capsule Endoscopy Delivery System
Acronym: RD-300
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: RD-300
Record Dates: First submitted 2010-03-15; First posted 2010-03-17 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Small Bowel Disease; Inflammatory Bowel Disease
Keywords: capsule endoscopy; small bowel disease; inflammatory bowel disease; Subjects indicated for EGD endoscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: To evaluate the safety and efficacy of an endoscopic capsule placement device.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PillCam® Express Capsule Endoscopy Delivery System — The PillCam® Express Capsule Endoscopy Delivery System is comprised of three parts: a catheter, a syringe and the capsule holder. The catheter is passed through the accessory channel of a standard endoscope and the capsule holder is snapped on to the distal end of the device. The endoscope is used to guide the Capsule Endoscopy Delivery System to the proximal duodenum. The capsule is then released pneumatically, using an air-filled syringe attached to the proximal end of the catheter.
  Once the capsule is deployed, the endoscope is withdrawn and the capsule holder is cut off at the distal part of the device with scissors. The catheter is then retracted and discarded.
  The PillCam® Express Capsule Endoscopy Delivery System is single-use, disposable and latex-free.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a trans-endoscopic capsule placement Capsule Endoscopy Delivery System.

DETAILED DESCRIPTION:
Natural ingestion of a wireless capsule endoscope (e.g. PillCam™ SB) is contraindicated in subjects with oropharyngeal or mechanical dysphagia, gastroparesis and known or suspected anatomical abnormalities. In addition, ingestion of a wireless capsule endoscope may be challenging in the pediatric population. The PillCam® Express Capsule Endoscopy Delivery System is intended to provide physicians with the capability to place capsules in the proximal duodenum using the accessory channel of a standard endoscope.

The PillCam™ SB capsule to be used in this study was cleared by the FDA in August 2001 for small bowel evaluation. It has been ingested to date by more than 1,000,000 people worldwide and is well accepted by subjects and physicians as well as the professional societies.

Further details of the PillCam®Express Capsule Endoscopy Delivery System can be found in the device description section.

This study is designed to evaluate the performance and safety of the Capsule Endoscopy Delivery System in subjects indicated to undergo a standard Esophagogastroduodenoscopy (EGD) endoscopy

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 2 years
* Subject scheduled for EGD endoscopy with a 2.8 mm (or greater) working channel

Exclusion criteria:

* Subject is known or is suspected to suffer from bowel obstruction or bowel perforation at the time of presentation
* Subject has history of UGI tract surgery (e.g., Billroth I, Billroth II, esophagectomy, gastrectomy, bariatric procedure)
* Presence of an electro-medical device (pacemaker or internal cardiac defibrillator)
* Subject is pregnant
* Subject is expected to undergo a MRI examination within 7 days after ingestion of the capsule
* Subject has known allergy to conscious sedation medications
* Subject or legal guardian is not able to provide written informed consent

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Leighton, MD, Principal Investigator — Mayo Clinic; Peter Legnani, MD, Principal Investigator — Private Practice New York, New York
Locations (3):
- United States (3):
  - Alabama Digestive Disorders Center, P. C., Huntsville, Alabama
  - Alabama Liver and Digestive Specialists, Montgomery, Alabama
  - RANY -Research Associates of New York (NY Gastroenterology Associates), New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 hospital sites
Groups:
- PillCam Express Capsule Delivery System: PillCam® Express Capsule Endoscopy Delivery System was used in conjunction with the endoscope to introduce a PillCam® SB capsule into the proximal duodenum. After the capsule was released in the designated location, a standard of care upper GI endoscopy was performed.
Period: Overall Study
Arm/Group | PillCam Express Capsule Delivery System
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PillCam Express Capsule Delivery System
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Capsule Placement Into the Duodenum Using Capsule Delivery System
Description: The number of capsules that successfully were in the duodenum as indicated by video images
Time Frame: up to 7 days
Measure: Number; unit: participants
Groups:
- Pillcam Express Capsule Delivery System: The delivery system is comprised of three parts: a catheter, a syringe and a capsule holder.
Arm/Group | Pillcam Express Capsule Delivery System
Number analyzed (Participants) | 25
participants | 25

2. Secondary Outcome: Physician's Subjective Assessment of the Ease of Capsule Placement
Description: The physician was required to assess the ease of use while answering a designated questionnaire.
  In addition, qualitative analysis was reformed with regard to all the open questions.
Time Frame: 7 days
Population: Physicians completed questionnaires for each of the 25 subjects. The questions were divided to two: physicians assessment A where 'YES' is associated with a smooth procedure (4 questions x 25 subjects = 100 Y/N assessments) and physicians B where 'no' is associated with smooth procedure (6 questions x 25 subjects = 150 Y/N assessment).
Measure: Number; unit: assessments
Units Other Than Participants: Y/N questions
Arm/Group | PillCam Express Capsule Delivery System
Number analyzed (Participants) | 25
Number analyzed (Y/N questions) | 250
assessments
  Physician Assessment A: number analyzed (Y/N questions) | 100
  Physician Assessment A | 94
  Physician Assessment B: number analyzed (Y/N questions) | 150
  Physician Assessment B | 126

ADVERSE EVENTS:
Time Frame: Adverse Event information was collected from screening (up to -14 day prior to procedure) through follow up phone contact at 5-10 days after the procedure
Arm/Group | PillCam Express Capsule Delivery System
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PillCam Express Capsule Delivery System (N=25)
capsule failed to deploy in first attempt (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No